CLINICAL TRIAL: NCT03613597
Title: A Randomized Phase II Trial of Etoposide Plus Lobaplatin Versus Etoposide Plus Cisplatin in Combination With Concurrent Thoracic Radiotherapy for Patients With Limited Small-cell Lung Cancer
Brief Title: Etoposide Plus Lobaplatin Versus Etoposide Plus Cisplatin for Patients With Limited Small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guizhou Medical University (Other)
Responsible Party: Principal Investigator, ShengFa Su, Professor, Guizhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-SCLC-001
Record Dates: First submitted 2018-07-22; First posted 2018-08-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; lobaplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoposide plus Lobaplatin group (Experimental): Chemotherapy:etoposide plus lobaplatin (EL)
  Interventions: Drug: etoposide plus lobaplatin
- Etoposide plus Cisplatin group (Active Comparator): Chemotherapy:etoposide plus cisplatin (EP)
  Interventions: Drug: etoposide plus cisplatin

INTERVENTIONS:
Drug: etoposide plus lobaplatin — Thoracic intensity modulated radiation therapy (IMRT) + etoposide plus lobaplatin
  Other Names: EL
  Arms: Etoposide plus Lobaplatin group
Drug: etoposide plus cisplatin — Thoracic intensity modulated radiation therapy (IMRT) + etoposide plus Cisplatin
  Other Names: EP
  Arms: Etoposide plus Cisplatin group

SUMMARY:
This randomized phase II study compare survival outcomes and toxicity of two chemotherapy regimens (etoposide plus lobaplatin or etoposide plus cisplatin) in combination with concurrent thoracic radiation therapy (TRT) for limited stage small cell lung cancer.

DETAILED DESCRIPTION:
Lobaplatin is a platinum complex with DNA alkylating activity that was developed by ASTA Medica (Degussa) for the treatment of cancer. Lobaplatin as the third-generation platinum antineoplastic agent, showed promising antineoplastic effects in variety of preclinical test tumor models. A randomized, multicenter phase III study showed that Lobaplatin plus etoposide (EL) regimen is not inferiority to cisplatin plus etoposide (EP) regimen in terms of PFS, the tolerance and QOL with EL regimen are better than that with EP regimen. Thus, we perform this study was to compare the efficacy and safety of EL and EP regimens concurrently with thoracic radiotherapy in patients with limited-stage SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed SCLC
* Newly diagnosed SCLC
* Either sex, age between 18 to 75 years
* Limited stage: AJCC (8th edition) Stage I-III (T any, N any, M0) that can be safely treated with definitive radiation doses. Excludes T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan.
* Performance status ECOG grade 0-1. Patients with PS 2 whose general condition is explained by obstructive/bulky disease likely to improve after the first cycle of chemotherapy can be included at the discretion of the local investigator. Patients with PS 2 as a result of comorbid conditions will be excluded.
* Adequate bone marrow, liver and renal function as defined below:neutrophils ≥ 1.5 × 109/L, platelets 80 × 109/L, hemoglobin ≥80 g/L, AST and ALT ≤2× the upper limit of the institutional normal range, total bilirubin ≤1.25× the upper limit of the institutional normal range, and creatinine concentration ≤120 μmol/L
* No history of thoracic surgery, radiation therapy, or chemotherapy
* Had measurable or assessable disease

Exclusion Criteria:

* Pregnancy or lactation at the time of enrollment
* Previous malignancy or other concomitant malignant disease
* Malignant pleural or pericardial effusions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | up to 12 months
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival(OS) | up to 24 months
  Overall survival is defined as the time interval from date of diagnosis to date of death from any cause
Treatment toxicities | up to 12 months
  To assess and record nausea, vomiting, hematologic toxicity,radiation oesophagitis and other treantment complications by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: ShengFa Su, PhD,MD, Principal Investigator — sushengfa2005@163.com
Locations (1):
- The affiliated hospital of Guizhou medical university, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang M, Ma Z, Li Q, Yang W, Chen X, Geng Y, Luo D, Hu Y, Wu B, Jiang W, Su S, Ouyang W, Lu B. Preliminary results of randomized phase II study of etoposide plus lobaplatin or etoposide plus cisplatin with concurrent thoracic radiotherapy in the treatment of limited-stage small cell lung cancer. Anticancer Drugs. 2023 Nov 1;34(10):1183-1189. doi: 10.1097/CAD.0000000000001501. Epub 2023 Jan 24. PMID 36727741